CLINICAL TRIAL: NCT00006116
Title: First Line Treatment of Stage IIIb/IV Non Small Cell (NSC) Lung Cancer With a Bimonthly Administration of a Combination of Cisplatin-Gemcitabine
Brief Title: Combination Chemotherapy in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068129; FRE-GERCOR-B98-1; EU-20026
Record Dates: First submitted 2000-08-03; First posted 2004-06-22 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2000-11

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining cisplatin with gemcitabine in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of the combination of cisplatin and gemcitabine in terms of response rate and progression free survival in patients with stage IIIB or IV non-small cell lung cancer. II. Evaluate this treatment regimen in terms of toxicity and quality of life in these patients.

OUTLINE: This is a multicenter study. Patients receive gemcitabine IV over 30 minutes and cisplatin IV over 1 hour every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients with no disease progression following 6 courses of therapy receive an additional 6 courses of therapy. Quality of life is assessed prior to each course and then every 3 months. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: A total of 37-83 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed non-small cell lung cancer Locally advanced Stage IIIB (T4, Nx, M0, or Tx, N3, M0) OR Metastatic disease Stage IV unresectable disease Following cell types eligible: Epidermoid cell Large cell Adenocarcinoma Bidimensionally measurable disease Unresectable recurrence after primary surgery allowed No brain metastasis

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: AST and ALT no greater than 3 times upper limit of normal (ULN) Bilirubin no greater than 1.5 times ULN Renal: Creatinine no greater than 1.10 mg/dL Cardiovascular: No uncontrolled cardiac disease Other: No other significant, uncontrolled underlying medical or psychiatric condition No serious active infection Neurologically stable No other prior malignancy except treated nonmelanomatous skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics Other: At least 30 days since prior experimental therapy No other concurrent experimental drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-04

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Terrioux, MD, Study Chair — Clinique de Docteur Terrioux
Locations (21):
- France (21):
  - Clinique Sainte Catherine, Avignon
  - C.H.G. Beauvais, Beauvais
  - Centre Hospitalier Departmental Felix Guyon, Bellepierre
  - Centre Hospitalier General, Brivé
  - Centre Hospitalier Emile Roux, Eaubonne
  - Centre Jean Bernard, Le Mans
  - C.H. Mans, Le Mans
  - Hopital Perpetuel Secours, Levallois-Perret
  - Clinique St. Faron, Mareuil-lès-Meaux
  - Clinique de Docteur Terrioux, Meaux
  - Clinique Hartmann, Neuilly-sur-Seine
  - American Hospital of Paris, Neuilly-sur-Seine
  - Clinique Du Mont Louis, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Hopital Claude Gallien, Quincy-sous-Sénart
  - Groupe Medical Saint Remy, Reims
  - Clinique les Bleuets, Reims
  - Polyclinique De Courlancy, Reims
  - Centre Rene Huguenin, Saint-Cloud
  - Centre du Rouget, Sarcelles